CLINICAL TRIAL: NCT05693441
Title: Study on the Chronic and Acute Effects of Nordic Berry Beverage on Cognitive Function, Cardiometabolic Risk Markers and Gut Microbiome: A Randomized, Double-blind, Placebo-controlled Intervention
Brief Title: Study on the Chronic and Acute Effects of Nordic Berry Beverage on Cognitive Function
Acronym: SCANBerry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aventure AB (Industry)
Collaborators: Berry Lab AB (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SCANBerry2022
Record Dates: First submitted 2022-11-17; First posted 2023-01-23 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Age-related Cognitive Decline
Keywords: cognitive function; memory

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active berry product (Active Comparator): Once daily consumption over the period of the study
  Interventions: Other: Active berry product
- Reference berry-like product (Placebo Comparator): Once daily consumption over the period of the study
  Interventions: Other: Reference berry-like product

INTERVENTIONS:
Other: Active berry product — Subjects should consume the active product containing nordic berries daily during the 12 week intervention period.
  Arms: Active berry product
Other: Reference berry-like product — Subjects should consume a reference product (isocaloric to active product, containing berry aromas and colouring but no actual berry compounds) daily during the 12 week intervention period.
  Other Names: Inactive control
  Arms: Reference berry-like product

SUMMARY:
The aim of the current study is to investigate whether acute and 12-weeks daily intake of Nordic berries can improve cognitive abilities of adults without cognitive disease, and whether the effect can be linked to changes in metabolic parameters.

DETAILED DESCRIPTION:
The study will be conducted with a randomized, double-blind, parallel-group (2 arms) placebo-controlled, single-center interventional design. The aim is to investigate the effects on cognitive function and cardiometabolic risk markers after acute and 12 weeks daily intake of a berry product vs. a reference product. The reference will be isocaloric and matched in taste, appearance, volume and macronutrient composition to the active berry product.

Two groups, each of 30 volunteers, are studied. One group of volunteers will consume the berry product while the other group act as control and will consume the reference product.

Each volunteer will be seen for a screening visit as well as one pre- and one post-intervention visit at the clinic. In addition, there will be 2 follow-up calls in between visits. Pre- and post intervention visits will include cognitive assessment with the CANTAB battery (episodic memory and verbal recognition memory), as well as additional cognitive and behavioral tests. Cardiometabolic parameters will be addressed (plasma glucose, insulin, inflammatory markers, blood lipids, body composition) and fecal samples collected.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60-85 years.
2. Capable and willing to give written informed consent.
3. Capable and willing to perform cognitive testing in Swedish (mastering the Swedish language, functional vision and hearing or the use of visual or hearing aids during testing).
4. Capable and willing to ingest the study beverage for 12 weeks and to follow the instructions given.
5. Agree to maintain consistent dietary habits and physical activity levels for the duration of the study

Exclusion Criteria:

1. Known to be affected by major neurocognitive disorder/dementia or low score on cognitive screening test (Mini Mental State Examination (MMSE) score less than 24.
2. Affected by other medical condition(s) or medication(s) known to significantly affect cognitive function.
3. Past history of brain damage, significant head trauma (including loss of consciousness as a result), brain surgery or stroke.
4. Underweight (BMI <18.5).
5. Significant psychiatric disorders with current symptoms.
6. Type 1 diabetes, recently diagnosis of Type 2 diabetes (<12 months) or ongoing insulin treatment.
7. Ongoing treatment for malignancy*.
8. Significant change in medication over the last 3 months.
9. Undergoing antibiotic therapy for the last 3 months prior to inclusion in the study.
10. Blood donation before (3 months) or during the study period.
11. Planned major intervention in health care or change in medication over the next 3 months (study period).
12. Currently active smoker or regular use of other nicotine products.
13. Drug or alcohol abuse.
14. Conditions with major impact on the gastrointestinal tract (such as Crohn's disease, ulcerative colitis, diagnosed gluten intolerance, undertaken intestinal resection or weight loss surgery).
15. Allergy / intolerance to berries or other ingredients in the study products (i.e., colorants, aromas, starch).
16. Vegetarians / vegans.
17. Daily, regular high consumption (approximately 1 dl or more per day) of berries or juices / marmalade / products with high content of bilberries and lingonberries. (Can be recruited if consumption has ceased to less than 5 grams of berries per day at least 1 month before visit 1.).
18. Taking supplements with potential cognitive effects (e.g., omega-3, ginko biloba, Souvenaid), or containing grape and berry extracts or probiotics (capsules or ProViva). (Can be recruited if this intake ceases at least one month before visit 1).
19. Planned longer absence/vacation during the next 3 months (study period).
20. Sharing household with someone participating in the current study
21. Concurrent participation in other clinical intervention trials (dietary/pharmacological).
22. Other reasons that make the SD in consultation with the PI deem the person inappropriate to include. *basalioma exempt from exclusion criteria

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Cognitive measures-memory | Change from baseline following 12 weeks daily consumption, compared to control
  Episodic memory - assessed using computerized cognitive battery including PAL (paired associates learning) test.
Cognitive measures-memory | Change from baseline following 12 weeks daily consumption, compared to control
  Episodic memory - assessed using computerized cognitive battery including VRM (verbal recognition memory) test
Cognitive measures - memory | Change from baseline at 1.5 hours post-dose, and 12 weeks daily consumption, compared to control
  Working memory - assessed using computerized cognitive battery including SWM (spatial working memory) test.
Cognitive measures - memory | Change from baseline at 1.5 hours post-dose, and 12 weeks daily consumption, compared to control
  Working memory - assessed using computerized cognitive battery including SDPT (symbol digits processing test).
Cognitive measures - executive function | Change from baseline at 1.5 hours post-dose, and 12 weeks daily consumption, compared to control
  Executive function - assessed using computerized cognitive battery including TMT (trail making test) A & B.
Cognitive measures - executive function | Change from baseline at 1.5 hours post-dose, and 12 weeks daily consumption, compared to control
  Executive function - assessed using computerized cognitive battery including PASAT (paced auditory serial addition test).
Cognitive measures - executive function | Change from baseline at 1.5 hours post-dose, and 12 weeks daily consumption, compared to control
  Executive function - assessed using computerized cognitive battery including Stroop test.
Cognitive measures - executive function | Change from baseline at 1.5 hours post-dose, and 12 weeks daily consumption, compared to control
  Executive function, verbal fluency - assessed using computerized cognitive battery including F-A-S test measuring word fluency
Cognitive measures - attention | Change from baseline at 1.5 hours post-dose, and 12 weeks daily consumption, compared to control
  Attention, reaction time - assessed using computerized cognitive battery including RTI (reaction time) test.
Cognitive measures | Change from baseline at 1.5 hours post-dose, and 12 weeks daily consumption, compared to control
  Global cognitive function - assessed by calculating a z-score from the cognitive battery score outcomes

SECONDARY OUTCOMES:
Circulating plasma biomarkers relating to cognitive function | Change from baseline at 1.5 hours post-dose, and 12 weeks daily consumption, compared to control
  Brain derived neurotrophic factor (BDNF)
Mood measurement | Change from baseline at 1.5 hours post-dose, and 12 weeks daily consumption, compared to control
  assessed using SCAS (the Swedish Core Affect Scale) mood questionnaire. A validated self-report measure of affective state. The SCAS comprises of 12 affective states that subjects rate on a scale from 1 - 10.
Self-reported quality of life | Difference from baseline vs control following 12 weeks of daily consumption
  assessed using the quality of life scale from the EQ-5D (EuroQol 5 Dimension) self-report survey. The subject grades their current overall quality of life on a scale 0-100.
Well-being measurement | Difference from baseline vs control following 12 weeks of daily consumption
  Assessed with World Health Organization- Five Well-Being Index (WHO-5). A validated 5 item scale for self-reporting levels of perceived well-being over the last two weeks. Items are rated using a 5-point scale.
Subjective memory | Difference from baseline vs control following 12 weeks of daily consumption
  Assessed using 3 simple questions about the subject's own memory evaluation. The subject is asked to rate their memory function (scale 0 to 7), how they percieve their own memory is working compared to others in the same age (0 to 5) and if anyone close to them has expressed concern over the subjects' memory
Cardiometabolic risk factor | Change from baseline at 1.5 hours post-dose, and 12 weeks daily consumption, compared to control
  blood pressure (SBP)
Cardiometabolic risk factor | Change from baseline at 1.5 hours post-dose, and 12 weeks daily consumption, compared to control
  blood pressure (DBP)
Cardiometabolic risk factor | Change from baseline at 1.5 hours post-dose, and 12 weeks daily consumption, compared to control
  Heart rate (HR)
Body composition | Change from baseline following 12 weeks daily consumption, compared to control
  Body weight (kg)
Body composition | Change from baseline following 12 weeks daily consumption, compared to control
  Body mass index (BMI) (e.g., weight (kg) and height (m) will be combined to report BMI in kg/m^2).
Body composition | Change from baseline following 12 weeks daily consumption, compared to control
  body fat % (measured by bioelectrical impedance analysis)
Body composition | Change from baseline following 12 weeks daily consumption, compared to control
  Waist circumference (cm)
Biomarkers of glycemia | Change from baseline at 1.5 hours post-dose, and 12 weeks daily consumption, compared to control
  glucose levels in blood
Biomarkers of glycemia | Change from baseline at 1.5 hours post-dose, and 12 weeks daily consumption, compared to control
  insulin levels in blood
Biomarkers of glycemia | Change from baseline following 12 weeks daily consumption, compared to control
  HOMA-IR (insulin resistance index, calculated based on fasting glucose and insulin levels)
Biomarkers of glycemia | Change from baseline following 12 weeks daily consumption, compared to control
  Fructosamine levels in blood
Biomarkers of lipemia in blood plasma | Difference from baseline vs control following 12 weeks of daily consumption
  triacylglycerols
Biomarkers of lipemia in blood plasma | Difference from baseline vs control following 12 weeks of daily consumption
  total cholesterol
Biomarkers of lipemia in blood plasma | Difference from baseline vs control following 12 weeks of daily consumption
  HDL-cholesterol
Biomarkers of lipemia in blood plasma | Difference from baseline vs control following 12 weeks of daily consumption
  LDL-cholesterol
Biomarkers of lipemia in blood plasma | Difference from baseline vs control following 12 weeks of daily consumption
  ApoB/A1
Biomarker endothelial function in blood plasma | Difference from baseline vs control following 12 weeks of daily consumption
  sVCAM-1
Biomarkers of liver function in blood plasma | Difference from baseline vs control following 12 weeks of daily consumption
  ALAT
Biomarkers of inflammation and oxidative stress blood plasma | Difference from baseline vs control following 12 weeks of daily consumption
  Interleukin
Biomarkers of inflammation and oxidative stress blood plasma | Difference from baseline vs control following 12 weeks of daily consumption
  acute phase proteins (C-reactive protein)

OTHER OUTCOMES:
Gut microbiota composition | Difference from baseline vs control following 12 weeks of daily consumption
  Sequencing of fecal samples
Gut function | Difference from baseline vs control following 12 weeks of daily consumption
  Questionnaire on gut function. The subject is asked to grade the frequency of symtomps of bloating, flatulence, abdominal pain and cramping, constipation and defecation pain, on a scale from 0 (never) to 3 (frequently).
Untargeted plasma metabolome | Difference from baseline vs control 1.5h post dose and following 12 weeks of daily consumption
  Untargeted plasma metabolomics will be employed to exploratively assess alterations in metabolites and to identify metabolites that increase or change with berry consumption
Explorative subgroup analyses (interactions) | Difference from baseline vs control 1.5h post dose and following 12 weeks of daily consumption
  Data analyses of how effects on the primary outcome (cognition) interacts with gender
Explorative subgroup analyses (interactions) | Difference from baseline vs control 1.5h post dose and following 12 weeks of daily consumption
  Data analyses of how effects on the primary outcome (cognition) interacts with age
Explorative subgroup analyses (interactions) | Difference from baseline vs control 1.5h post dose and following 12 weeks of daily consumption
  Data analyses of how effects on the primary outcome (cognition) interacts with sex
Explorative subgroup analyses (interactions) | Difference from baseline vs control 1.5h post dose and following 12 weeks of daily consumption
  Data analyses of how effects on the primary outcome (cognition) interacts with dietary habits
Explorative subgroup analyses (interactions) | Difference from baseline vs control 1.5h post dose and following 12 weeks of daily consumption
  Data analyses of how effects on the primary outcome (cognition) interacts with education level
Explorative subgroup analyses (interactions) | Difference from baseline vs control 1.5h post dose and following 12 weeks of daily consumption
  Data analyses of how effects on the primary outcome (cognition) interacts with intake of permitted medications
Adverse events | Through study completion (12 weeks)
  Unexpected health problems and safety outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Aventure AB, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No